CLINICAL TRIAL: NCT04241965
Title: A Phase 1b, Single-blind, Placebo-controlled, Adaptive Design, Outpatient Trial to Assess the Effects of Single Oral Tablet Doses of OPC-214870 on Photic-induced Paroxysmal Electroencephalogram Responses in Subjects Who Have Demonstrated Photoepileptiform Discharges on Electroencephalogram With or Without Seizures
Brief Title: A Single-blind, Placebo-controlled, Outpatient Trial to Assess the Effects of Single Oral Tablet Dose of OPC-214870
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 325-201-00003
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention 1 (Experimental): Single dose; up to 400 mg capsule; adaptive dosage determined by initial dosing from cohort 1.Potential for a matching placebo dose to be administered.
  Interventions: Drug: OPC-214870; Other: Placebo
- Placebo (Placebo Comparator): Single dose; potential for a matching OPC-214870 dose to be administered.
  Interventions: Drug: OPC-214870; Other: Placebo

INTERVENTIONS:
Drug: OPC-214870 — Tablet(s)
Other: Placebo — Tablet(s)

SUMMARY:
Despite availability of several antiepileptic drugs (AEDs), in one-third of patients, epilepsy remains uncontrolled with AEDs. There is a need to develop new approaches to improve the existing medications to relieve patients' epilepsy, and OPC-214870 is being studied for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 and 64 years of age, inclusive.
* Body mass index (BMI) between 18 and 40 kg/m^2, inclusive.
* Subjects with a diagnosis and history of photoparoxysmal response on EEG.
* Subjects must be stable for 1 month prior to screening. Stable is defined as having no change in concomitant therapy and no worsening in the opinion of the investigator.
* Subjects may be treatment-naïve to AEDs or currently treated with up to 3 AEDs.
* Subjects must have a reproducible standardized photosensitivity range on EEG of at least 3 points in at least 1 eye condition.
* Subjects who agree to remain abstinent, or practice double-barrier forms of birth control, from trial to screening through 90 days after the last dose of IMP, OR males and females of non-childbearing potential who are documented as sterile (i.e. male subjects who have undergone bilateral orchidectomy and female subjects who have undergone bilateral oophorectomy, bilateral salpingectomy, or hysterectomy, or who have been postmenopausal for at least 12 months.

Exclusion Criteria:

* History of non-epileptic seizures
* History of status epilepticus in the past 5 years
* An active central nervous system (CNS) infection, demyelinating disease, degenerative neurological disease, or any CNS disease deemed to be progressive during the course of the trial that may confound the interpretation of the trial results.
* Positive urine drug screen for substance of abuse or upon check in to the trial site. Benzodiazepines are excluded as a drug of abuse, but are allowed as rescue medication or when part of subject's stable concomitant medication at enrollment.
* History of drug and/or alcohol abuse within 24 months prior to screening.
* Consumption of grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 7 days prior to dosing.
* Consumption of more than 1 alcoholic drink within 24 hours prior to dosing. Food and beverages containing methylxanthines (caffeinated coffee, caffeinated tea, caffeinated soda, and chocolate) must remain stable throughout the trial.
* Extreme physical activity within 24 hours before screening and visit
* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP
* Subject having taken an investigational drug within 30 days preceding screening.
* Use of over-the-counter drugs, herbal medicines, or vitamin supplements within 14 days or 5 half-lives, whichever is longer, prior to dosing and antibiotics within 30 days prior to dosing.
* Subjects who had neurosurgery in last 6 months.
* Subjects on a ketogenic diet.
* History of significant sleep disorders, or any disorder or activity that causes sleep deprivation.
* Subjects who work "night shifts"
* Subjects with uncontrolled sleep disorders; subjects should be on a stable dose of sleep medications.
* History of, or current hepatitis or acquired immunodeficiency syndrome or carriers of hepatitis B surface antigen (HBsAg), hepatitis C antibodies (anti-HCV), and/or HIV antibodies.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Change in Standardized Photosensitivity Range (SPR) | Up to 3 days
  OPC-214870 in comparison to placebo

SECONDARY OUTCOMES:
Onset and duration of SPR | Up to 3 days
  OPC-214870 in comparison to placebo

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Ormond Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com